CLINICAL TRIAL: NCT04025281
Title: Post-prandial Effects of Extra Virgin Olive Oil on Endothelial Function in Adults at Risk for Type 2 Diabetes: A Randomized Crossover Controlled Trial
Brief Title: Post-prandial Effects of Extra Virgin Olive Oil on Endothelial Function in Adults at Risk for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffin Hospital (Other)
Responsible Party: Principal Investigator, VALENTINE NJIKE, PRINCIPAL INVESTIGATOR, Griffin Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2018-12
Record Dates: First submitted 2019-07-17; First posted 2019-07-18 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: To provide a sound basis for the statistical comparison of outcome measures for treatment assignments, participants will be randomized to 1 of 2 sequence permutations of extra virgin olive oil enriched meal and refined olive oil enriched meal. Each permutation will include a first treatment assignment, followed by a 1-week washout phase, and followed by a second treatment assignment.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extra virgin olive oil (Active Comparator): Participants will consume a meal prepared with 50 mL extra virgin olive oil. The meals will be prepared and provided to the study participants in the cafeteria of Griffin Hospital, where the Prevention Research Center is located. With the exception of the type of olive oil used in the meals, the meal plan will be comparable in all the intervention phases for the same individual.
  Interventions: Other: Extra Virgin Olive Oil
- Refined olive oil (Active Comparator): Participants will consume a meal prepared with 50 mL refined olive oil in the cafeteria of Griffin Hospital. With the exception of the olive oil used, the meal plan will be comparable in each the intervention phases for the same individual.
  Interventions: Other: Refined Olive Oil

INTERVENTIONS:
Other: Extra Virgin Olive Oil — Participants will consume a meal prepared with 50 mL extra virgin olive oil. The meals will be prepared and provided to the study participants in the cafeteria of Griffin Hospital, where the Prevention Research Center is located. With the exception of the type of olive oil used in the meals, the meal plan will be comparable in all the intervention phases for the same individual.
  Arms: Extra virgin olive oil
Other: Refined Olive Oil — Participants will consume a meal prepared with 50 mL refined olive oil in the cafeteria of Griffin Hospital. With the exception of the olive oil used, the meal plan will be comparable in each the intervention phases for the same individual.
  Arms: Refined olive oil

SUMMARY:
Purpose:

The number of cases of adults with Type 2 diabetes has quadrupled since 1980. This increase in the number of cases of diabetes is attributed to changes in dietary patterns, which include an increase in the consumption of obesogenic foods such as sugary foods and beverages. Patients with diabetes or at risk for diabetes are more likely to develop a cardiovascular event. Though glycemic control remains the basis of diabetes care, the co-management of atherosclerosis, hypertension and cardiovascular risk reduction, and prevention of long-term consequences are also important predictable measures to improve survival. The progression from prediabetes to Type 2 diabetes and complications of diabetes could be prevented. Lifestyle interventions (i.e., nutrition and physical activity) are the cornerstone for the primary prevention of Type 2 diabetes. Healthful eating can also improve cardio-metabolic risk factors associated with those at risk for or Type 2 diabetes. Foods that are low in fat and calories and high in fiber, with a focus on fruit, vegetables, whole grains, and the inclusion of healthful oils in their diets are typically recommended to prevent the progression from prediabetes to diabetes and complications of diabetes. Diets rich in mono- and polyunsaturated fatty acids have been shown to improve cardio-metabolic health in those at risk for or with Type 2 diabetes patients. However, the effect of olive oils on endothelial function (a surrogate marker of cardiovascular risk) in adults at risk for Type 2 diabetes is controversial. Refined olive oils lack important antioxidants and anti-inflammatory properties. Extra virgin olive oils have relatively higher levels of some minor phenolic compounds, and more naturally-occurring minerals and vitamins found in olives, that are essential to improve cardio-metabolic risk factors in those at risk for or with Type 2 diabetes. We propose a prospective, randomized, controlled crossover study to assess the post-prandial effects of extra virgin olive oil, versus post-prandial effects of a refined olive oil, on endothelial function and blood pressure in adults at risk for Type 2 diabetes.

Specific Aims To assess the post-prandial effect of extra virgin olive oil on endothelial function, measured as flow mediated dilatation, in adults at risk for Type 2 diabetes. Specifically, to demonstrate at least a 3.5% improvement in endothelial function following the consumption of a meal with 50 mL of extra virgin olive oil, compared with a meal with 50 mL of refined olive oil, in individuals at risk for Type 2 diabetes.

To assess the post-prandial effect of extra virgin olive oil on blood pressure in adults at risk for Type 2 diabetes. Specifically, to demonstrate at least 3 mmHg improvements in systolic and diastolic blood pressure after the consumption of a meal with 50 mL of extra virgin olive oil compared with a meal with 50 mL of refined olive oil, in individuals at risk for Type 2 diabetes.

Hypotheses Consumption of a meal with extra virgin olive oil compared with a meal with refined olive oil will show superior benefits in endothelial function in adults at risk for Type 2 diabetes.

Consumption of a meal with extra virgin olive oil compared with a meal with refined olive oil will show better improvement in blood pressure in adults at risk for Type 2 diabetes.

DETAILED DESCRIPTION:
Diabetes is a public health problem of epidemic proportions. According to the 2017 National Diabetes Statistics Report, 30 million people, or 9.4% of the U.S. population, are estimated to have diabetes, of which 23.1 million people are diagnosed. About 84.1 million people, or 1 in 3 people in the U.S., are estimated to have prediabetes, yet only 1 out 10 people with prediabetes is aware that they have this condition. Of those with prediabetes, 15-30% are likely to develop Type 2 diabetes within 5 years. The total medical costs and lost work and wages for people with diagnosed diabetes is about $245 billion, with the medical costs for people with diabetes being twice as high as for those without diabetes. The risk of death in individuals with diabetes is more than 50% higher than for adults without diabetes. Type 2 diabetes accounts for about 90% to 95% of all diagnosed cases of diabetes. Diabetes is the seventh leading cause of death in the U.S. Diabetes complications include cardiovascular disease (CVD), stroke, hypertension, blindness, kidney disease, nervous system damage, limb amputations, and biochemical imbalances that can cause acute life-threatening events. Rates of cardiovascular mortality are 2 to 4 times higher among adults with diabetes than among those without diabetes.

Epidemiological and cohort studies show a clear and consistent correlation of hyperglycemia with CVD. High glucose activates a pro-atherogenic phenotype in the vessel wall of endothelial cells, vascular smooth muscle cells, inflammatory cells, fibroblasts, and platelets, leading to a feed-forward atherogenic response. Diets with a low glycemic load have been reported to improve serum lipid profiles, reduce C-reactive protein (CRP) levels, and aid in weight control. In cross-sectional studies, they have been associated with higher levels of high-density lipoprotein cholesterol (HDL-C), with reduced CRP concentrations, and, in cohort studies, with decreased risk of developing diabetes and CVD. Insulin resistance may also contribute to high blood pressure, increased triglycerides and LDL cholesterol, and reduced levels of HDL cholesterol. While glycemic control remains a cornerstone of diabetes care, the co-management of hypertension, atherosclerosis, cardiovascular risk reduction, and prevention of long-term consequences are also recognized as essential to improve long-term survival.

The cornerstone of the management and prevention of Type 2 diabetes is lifestyle intervention. Prior studies have shown an association between improvement in cardio-metabolic health and diets rich in olive oils. Low glycemic index foods are typically recommended for patients with Type 2 diabetes or at risk for Type 2 diabetes. Extra virgin olive oil is a nutrient-dense food with a low glycemic index. It is rich in mono-unsaturated fatty acids that are vital to improve cardio-metabolic risk factors in those at risk for Type 2 diabetes. Among all the oils, olive oils have a relatively high content of monounsaturated fatty acids. Diets rich in mono- and polyunsaturated fatty acids have shown favorable effects on cardiovascular health, glycemic control, insulin sensitivity, and lipid profile. All olive oils, (inclusive of extra virgin olive oil), have a relatively higher amount of monounsaturated fatty acids. While refined olive oils lack important antioxidants and anti-inflammatory properties, extra virgin olive oils specifically contains relatively higher levels of some minor phenolic compounds, along with more naturally-occurring minerals and vitamins found in olives that have favorable effects on cardio-metabolic health. Therefore, the inclusion of extra virgin olive oil in the diets of adults at risk for Type 2 diabetes is likely to confer better cardio-metabolic health benefits than a refined olive oil. Some oils improve, and some impair, endothelial function. Published studies have said both about olive oils, probably because the status and caliber of the olive oils was not always specified. We therefore propose to differentiate 'good' from 'bad' olive oils, and to show that extra virgin olive oils have decisively beneficial effects, while those effects are attenuated or lost as the oil is degraded. Specifically, proposed is a randomized crossover controlled trial to assess the impact of extra virgin olive oil, as compared with refined olive oil, on endothelial function in adults at risk for Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female age 25-75 years;
2. non-smokers;
3. post-menopausal females not currently on hormone replacement therapy;
4. at risk for Type 2 diabetes as defined by meeting at least one of the criteria listed below: (a) metabolic syndrome, i.e. meet 3 out of 5 of the following criteria: (i) blood pressure >130/85 mmHg or currently taking antihypertensive medication; (ii) fasting plasma glucose (FPG) >100 mg/dL (6.1 mmol/L); (iii) serum triglycerides level (TG)>150 mg/dL (1.69 mmol/L); (iv) high-density lipoprotein (HDL) cholesterol < 40 mg/dL (1.04 mmol/L) in men, and < 50 mg/dL (1.29 mmol/L) in women; (v) overweight (body mass index, or BMI ≥25kg/m²) with waist circumference of more than 40 inches (102 cm) for men and more than 35 inches (88 cm) for women; (b) fasting blood glucose >100mg/dL and <126mg/dL or hemoglobin A1C 5.7-6.4 %.

Exclusion Criteria:

1. failure to meet inclusion criteria;
2. anticipated inability to complete study protocol for any reason;
3. current eating disorder;
4. use of insulin, glucose-sensitizing medication, vasoactive medication (including glucocorticoids, antineoplastic agents, psychoactive agents, or bronchodilators) or nutraceuticals;
5. regular use of fiber supplements;
6. diabetes;
7. sleep apnea;
8. restricted diets by choice (e.g., vegetarian, vegan);
9. coagulopathy, known bleeding diathesis, or history of clinically significant hemorrhage, or current use of warfarin;
10. regular exercise as defined by participating in moderate-intensity > 150 minutes/week.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Endothelial Function (EF) Assessment | 2 hours
  Endothelial function will be measured as Flow-mediated dilatation (FMD), that is the percent change in brachial artery diameter from pre-cuff inflation to 60-seconds post-cuff release. In addition to brachial diameter at 60 seconds post-cuff release, flow after cuff deflation within the first 15 seconds will be used as an indicator of stimulus strength, hyperemic flow being the stimulus for endothelial reactivity. To account for potential variability in stimulus strength, a secondary analysis will be performed in which FMD is divided by flow at 15 seconds post-cuff deflation to create a stimulus-adjusted response measure.

SECONDARY OUTCOMES:
Office Blood Pressure | 2 hours
  Systolic and diastolic BP will be measured at each visit using an approved automated device. Blood pressure will be measured (average of two measurements with five minutes between measurements) with the participant sitting in a quiet room.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-Griffin Prevention Research Center, Derby, Connecticut, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention. National Diabetes Statistics Report.2017. https://www.cdc.gov/diabetes/pdfs/data/statistics/national-diabetes-statistics-report.pdf. Accessed 09/11/2018
- [Background] Centers for Disease Control and Prevention. National diabetes fact sheet: national estimates and general information on diabetes and prediabetes in the United States, 2011. Available from: http://www.cdc.gov/diabetes/pubs/pdf/ndfs_2011.pdf. Accessed 09/11/2018
- [Background] Reusch JE, Wang CC. Cardiovascular disease in diabetes: where does glucose fit in? J Clin Endocrinol Metab. 2011 Aug;96(8):2367-76. doi: 10.1210/jc.2010-3011. Epub 2011 May 18. PMID 21593112
- [Background] Esfahani A, Wong JM, Mirrahimi A, Srichaikul K, Jenkins DJ, Kendall CW. The glycemic index: physiological significance. J Am Coll Nutr. 2009 Aug;28 Suppl:439S-445S. doi: 10.1080/07315724.2009.10718109. PMID 20234030
- [Background] Bitzur R, Cohen H, Kamari Y, Shaish A, Harats D. Triglycerides and HDL cholesterol: stars or second leads in diabetes? Diabetes Care. 2009 Nov;32 Suppl 2(Suppl 2):S373-7. doi: 10.2337/dc09-S343. No abstract available. PMID 19875584
- [Background] Casas R, Sacanella E, Urpi-Sarda M, Chiva-Blanch G, Ros E, Martinez-Gonzalez MA, Covas MI; Rosa Ma Lamuela-Raventos; Salas-Salvado J, Fiol M, Aros F, Estruch R. The effects of the mediterranean diet on biomarkers of vascular wall inflammation and plaque vulnerability in subjects with high risk for cardiovascular disease. A randomized trial. PLoS One. 2014 Jun 12;9(6):e100084. doi: 10.1371/journal.pone.0100084. eCollection 2014. PMID 24925270
- [Background] Pedret A, Fernandez-Castillejo S, Valls RM, Catalan U, Rubio L, Romeu M, Macia A, Lopez de Las Hazas MC, Farras M, Giralt M, Mosele JI, Martin-Pelaez S, Remaley AT, Covas MI, Fito M, Motilva MJ, Sola R. Cardiovascular Benefits of Phenol-Enriched Virgin Olive Oils: New Insights from the Virgin Olive Oil and HDL Functionality (VOHF) Study. Mol Nutr Food Res. 2018 Aug;62(16):e1800456. doi: 10.1002/mnfr.201800456. Epub 2018 Jul 30. PMID 29956886
- [Background] Martin-Pelaez S, Mosele JI, Pizarro N, Farras M, de la Torre R, Subirana I, Perez-Cano FJ, Castaner O, Sola R, Fernandez-Castillejo S, Heredia S, Farre M, Motilva MJ, Fito M. Effect of virgin olive oil and thyme phenolic compounds on blood lipid profile: implications of human gut microbiota. Eur J Nutr. 2017 Feb;56(1):119-131. doi: 10.1007/s00394-015-1063-2. Epub 2015 Nov 5. PMID 26541328
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary prevention of cardiovascular disease with a Mediterranean diet. N Engl J Med. 2013 Apr 4;368(14):1279-90. doi: 10.1056/NEJMoa1200303. Epub 2013 Feb 25. PMID 23432189 (Retraction: PMID 29897867 N Engl J Med. 2018 Jun 21;378(25):2441-2442)
- [Background] George ES, Marshall S, Mayr HL, Trakman GL, Tatucu-Babet OA, Lassemillante AM, Bramley A, Reddy AJ, Forsyth A, Tierney AC, Thomas CJ, Itsiopoulos C, Marx W. The effect of high-polyphenol extra virgin olive oil on cardiovascular risk factors: A systematic review and meta-analysis. Crit Rev Food Sci Nutr. 2019;59(17):2772-2795. doi: 10.1080/10408398.2018.1470491. Epub 2018 Nov 13. PMID 29708409
- [Background] Arpon A, Milagro FI, Razquin C, Corella D, Estruch R, Fito M, Marti A, Martinez-Gonzalez MA, Ros E, Salas-Salvado J, Riezu-Boj JI, Martinez JA. Impact of Consuming Extra-Virgin Olive Oil or Nuts within a Mediterranean Diet on DNA Methylation in Peripheral White Blood Cells within the PREDIMED-Navarra Randomized Controlled Trial: A Role for Dietary Lipids. Nutrients. 2017 Dec 23;10(1):15. doi: 10.3390/nu10010015. PMID 29295516
- [Background] Mensink RP, Katan MB. Effect of monounsaturated fatty acids versus complex carbohydrates on high-density lipoproteins in healthy men and women. Lancet. 1987 Jan 17;1(8525):122-5. doi: 10.1016/s0140-6736(87)91965-9. PMID 2879969
- [Background] Grundy SM, Florentin L, Nix D, Whelan MF. Comparison of monounsaturated fatty acids and carbohydrates for reducing raised levels of plasma cholesterol in man. Am J Clin Nutr. 1988 Jun;47(6):965-9. doi: 10.1093/ajcn/47.6.965. PMID 3376911
- [Background] Fulgoni VL 3rd, Dreher M, Davenport AJ. Avocado consumption is associated with better diet quality and nutrient intake, and lower metabolic syndrome risk in US adults: results from the National Health and Nutrition Examination Survey (NHANES) 2001-2008. Nutr J. 2013 Jan 2;12:1. doi: 10.1186/1475-2891-12-1. PMID 23282226
- [Background] Franz MJ, Horton ES Sr, Bantle JP, Beebe CA, Brunzell JD, Coulston AM, Henry RR, Hoogwerf BJ, Stacpoole PW. Nutrition principles for the management of diabetes and related complications. Diabetes Care. 1994 May;17(5):490-518. doi: 10.2337/diacare.17.5.490. No abstract available. PMID 8062628
- [Background] Nutritional Recommendations and Principles for People with Diabetes Mellitus. Diabetes Care. 1998;21(S-1):S32-S35.
- [Background] Rueda-Clausen CF, Silva FA, Lindarte MA, Villa-Roel C, Gomez E, Gutierrez R, Cure-Cure C, Lopez-Jaramillo P. Olive, soybean and palm oils intake have a similar acute detrimental effect over the endothelial function in healthy young subjects. Nutr Metab Cardiovasc Dis. 2007 Jan;17(1):50-7. doi: 10.1016/j.numecd.2005.08.008. Epub 2006 Mar 20. PMID 17174226
- [Background] Sanchez-Rodriguez E, Lima-Cabello E, Biel-Glesson S, Fernandez-Navarro JR, Calleja MA, Roca M, Espejo-Calvo JA, Gil-Extremera B, Soria-Florido M, de la Torre R, Fito M, Covas MI, Alche JD, Martinez de Victoria E, Gil A, Mesa MD. Effects of Virgin Olive Oils Differing in Their Bioactive Compound Contents on Metabolic Syndrome and Endothelial Functional Risk Biomarkers in Healthy Adults: A Randomized Double-Blind Controlled Trial. Nutrients. 2018 May 16;10(5):626. doi: 10.3390/nu10050626. PMID 29772657
- [Background] Torres-Pena JD, Garcia-Rios A, Delgado-Casado N, Gomez-Luna P, Alcala-Diaz JF, Yubero-Serrano EM, Gomez-Delgado F, Leon-Acuna A, Lopez-Moreno J, Camargo A, Tinahones FJ, Delgado-Lista J, Ordovas JM, Perez-Martinez P, Lopez-Miranda J. Mediterranean diet improves endothelial function in patients with diabetes and prediabetes: A report from the CORDIOPREV study. Atherosclerosis. 2018 Feb;269:50-56. doi: 10.1016/j.atherosclerosis.2017.12.012. Epub 2017 Dec 8. PMID 29274507
- [Background] Davis CR, Hodgson JM, Woodman R, Bryan J, Wilson C, Murphy KJ. A Mediterranean diet lowers blood pressure and improves endothelial function: results from the MedLey randomized intervention trial. Am J Clin Nutr. 2017 Jun;105(6):1305-1313. doi: 10.3945/ajcn.116.146803. Epub 2017 Apr 19. PMID 28424187
- [Background] Storniolo CE, Casillas R, Bullo M, Castaner O, Ros E, Saez GT, Toledo E, Estruch R, Ruiz-Gutierrez V, Fito M, Martinez-Gonzalez MA, Salas-Salvado J, Mitjavila MT, Moreno JJ. A Mediterranean diet supplemented with extra virgin olive oil or nuts improves endothelial markers involved in blood pressure control in hypertensive women. Eur J Nutr. 2017 Feb;56(1):89-97. doi: 10.1007/s00394-015-1060-5. Epub 2015 Oct 8. PMID 26450601
- [Background] Njike VY, Yarandi N, Petraro P, Ayettey RG, Treu JA, Katz DL. Inclusion of walnut in the diets of adults at risk for type 2 diabetes and their dietary pattern changes: a randomized, controlled, cross-over trial. BMJ Open Diabetes Res Care. 2016 Oct 19;4(1):e000293. doi: 10.1136/bmjdrc-2016-000293. eCollection 2016. PMID 27843557
- [Background] Njike VY, Ayettey R, Petraro P, Treu JA, Katz DL. Walnut ingestion in adults at risk for diabetes: effects on body composition, diet quality, and cardiac risk measures. BMJ Open Diabetes Res Care. 2015 Oct 19;3(1):e000115. doi: 10.1136/bmjdrc-2015-000115. eCollection 2015. PMID 26688734
- [Background] Ma Y, Njike VY, Millet J, Dutta S, Doughty K, Treu JA, Katz DL. Effects of walnut consumption on endothelial function in type 2 diabetic subjects: a randomized controlled crossover trial. Diabetes Care. 2010 Feb;33(2):227-32. doi: 10.2337/dc09-1156. Epub 2009 Oct 30. PMID 19880586
- [Background] Katz DL, Davidhi A, Ma Y, Kavak Y, Bifulco L, Njike VY. Effects of walnuts on endothelial function in overweight adults with visceral obesity: a randomized, controlled, crossover trial. J Am Coll Nutr. 2012 Dec;31(6):415-23. doi: 10.1080/07315724.2012.10720468. PMID 23756586
- [Background] Njike VY, Kavak Y, Treu JA, Doughty K, Katz DL. Snacking, Satiety, and Weight: A Randomized, Controlled Trial. Am J Health Promot. 2017 Jul;31(4):296-301. doi: 10.4278/ajhp.150120-QUAN-676. Epub 2015 Nov 11. PMID 26559707
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Derived] Njike VY, Ayettey R, Treu JA, Doughty KN, Katz DL. Post-prandial effects of high-polyphenolic extra virgin olive oil on endothelial function in adults at risk for type 2 diabetes: A randomized controlled crossover trial. Int J Cardiol. 2021 May 1;330:171-176. doi: 10.1016/j.ijcard.2021.01.062. Epub 2021 Feb 3. PMID 33548380